CLINICAL TRIAL: NCT02923934
Title: A Phase II Clinical Trial Evaluating Ipilimumab and Nivolumab in Combination for the Treatment of Rare Gastrointestinal, Neuro-Endocrine and Gynaecological Cancers
Brief Title: A Phase II Trial of Ipilimumab and Nivolumab for the Treatment of Rare Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONJ2016-001
Record Dates: First submitted 2016-10-02; First posted 2016-10-05 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Gastrointestinal Cancer; Neuroendocrine Tumours; Malignant Female Reproductive System Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neuroendocrine Tumors | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Masking Description: This is an open label study, all patients receive the same treatment as per the protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ipilimumab and Nivolumab (Experimental): All Subjects will be treated with: Nivolumab at 3 mg/kg and ipilimumab at 1 mg/kg concurrently every 3 weeks for 4 doses followed by nivolumab only at 3mg/kg every 2 weeks until progression (up to 48 total doses of nivolumab)
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) is a key regulator of T cell activity. Ipilimumab is a CTLA-4 immune checkpoint inhibitor that blocks T-cell inhibitory signals induced by the CTLA-4 pathway, increasing the number of tumor reactive T effector cells which mobilize to mount a direct T-cell immune attack against tumor cells. CTLA-4 blockade can also reduce T regulatory cell function, which may lead to an increase in anti-tumor immune response.
  Other Names: YERVOY ®
Drug: Nivolumab — A fully human immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed cell death-1 (PD-1,PCD-1) with immune checkpoint inhibitory and antineoplastic activities. Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs (antigen presenting cells). This results in the activation of T-cells and cell-mediated immune responses against tumor cells or pathogens. Activated PD-1 negatively regulates T-cell activation and and plays a key role in in tumor evasion from host immunity.
  Other Names: Opdivo

SUMMARY:
The three tumour streams that will be studied in this protocol are: (i) upper GI malignancies (comprising intra-hepatic/extra-hepatic cholangiocarcinomas,gall bladder cancers and duodenal cancers).); (ii) neuroendocrine tumours (inc. Pancreatic, bronchial and intestinal carcinoid tumours) and (iii) rare gynaecological tumours (including but will not be limited to: vaginal or vulval carcinomas, clear cell carcinoma of the ovary, low grade serous ovarian cancer, mixed mullarian tumours (carcinosarcoma), sarcomas of the female genital tract and granulosa cell tumours).

The role of immunotherapy is being defined in more common cancer types, however because of their rarity, the efficacy of immunotherapy for these cancers is poorly defined.

This protocol provides an important opportunity to establish whether the combination of nivolumab & ipilimumab has efficacy in these cancers.

DETAILED DESCRIPTION:
This is a phase 2 clinical trial of nivolumab combined with ipilimumab in subjects with rare cancers. This study will allow an evaluation of the clinical benefit, as measured by progression free survival (PFS) and overall survival (OS), provided by nivolumab combined with ipilimumab. If the safety profile is acceptable and clinically efficacy is seen, this study would support the use of nivolumab combined with ipilimumab in subjects with these cancers.

Study Rationale Clinically advanced rare cancers pose a significant clinical challenge because evidence based treatments are seldom available for patients suffering from these malignancies. Despite little evidence that shows clinical benefit, these patients are often treated with chemotherapeutic agents that are used in patients with more common malignancies that arise from the same anatomical site. Furthermore, because of small numbers, they are often excluded from clinical trials with newer agents. The rare care project has defined a rare malignancy as a cancer with an incidence of less than 6/100000/year. It is estimated that 42,000 people are diagnosed with a form of rare or less common cancer in Australia every year (www.canceraustralia.gov.au). The cancer specific survival of patients diagnosed with a rare malignancy is significantly lower than with common cancers highlighting the need to improve management and treatment of these patients. Given the recent success of cancer immunotherapy with checkpoint regulators such as ipilimumab and nivolumab in a whole range of different cancer types, it can be postulated that these agents could be beneficial in rare cancers and improve the overall outlook of patients with these conditions. It is proposed here that patient cohorts which fall within three distinct tumour streams will be examined, with all patients receiving ipilimumab and nivolumab as combination immunotherapy. The three tumour streams are defined as: upper GI malignancies (comprising intra-hepatic/ extra-hepatic cholangiocarcinomas,gall bladder cancers and duodenal cancers).); neuroendocrine tumours (inc. Pancreatic, bronchial and intestinal carcinoid tumours) and rare gynaecological tumours (including but will not be limited to: vaginal or vulval carcinomas, clear cell carcinoma of the ovary, low grade serous ovarian cancer, mixed mullarian tumours (carcinosarcoma), sarcomas of the female genital tract and granulosa cell tumours). Although overall response rates for individual tumour types will not be established due to sample size (target 20 patients per tumour stream, n=60 total), descriptive information of individual patient responses will guide immune-directed therapies to responsive rare tumour types and may be broadened to tumour streams.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
2. Target Population

   * Histologically confirmed Upper GI malignancies (Cholangiocarcinoma/ duodenal carcinoma - collect MSI (microsatellite instability) status); Neuroendocrine tumours (inc. pancreatic, bronchial and intestinal carcinoid tumours) and Rare Gynaecological tumours (including but will not be limited to: vaginal or vulval carcinomas, clear cell carcinoma of the ovary, low grade serous ovarian cancer, mixed Mullarian tumours (carcinosarcoma), sarcomas of the female genital tract and granulosa cell tumours).
   * Eastern Cooperative Oncology Group (ECOG) performance status of 1
   * Prior systemic therapy is permitted if it was completed at least 4 weeks prior to enrolment, and all related adverse events have either returned to baseline or stabilized or subjects are not suitable for, or if declining established standard therapies.
   * Prior radiotherapy must have been completed at least 2 weeks prior to study drug administration.
   * Measurable disease by CT or MRI per RECIST 1.1 criteria
   * Tumour tissue from an unresectable or metastatic site of disease must be provided for biomarker analyses. If an insufficient amount of tumour tissue from an unresectable or metastatic site is available prior to the start of the screening phase, subjects must consent to allow the acquisition of additional tumour tissue for performance of biomarker analyses.
   * Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization:

     * WBC (white blood cells) > or = to 2000/μL
     * Neutrophils > or = to 1500/μL
     * Platelets > or = to 100 x103/μL
     * Hemoglobin > 9.0 g/dL
     * Serum creatinine < or = to 1.5 x ULN or creatinine clearance (CrCl) 40 mL/min (using the Cockcroft-Gault formula)
     * AST/ALT (aspartate transaminase/alanine transaminase) < or = to 3 x ULN
     * Total Bilirubin < or = to 1.5 x ULN (Upper limit of normal) (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL).
   * Subject Re-enrolment: This study permits the re-enrolment of a subject that has discontinued the study as a pre-treatment failure (i.e. subject has not been treated) after obtaining agreement from the medical monitor prior to re enrolling a subject. If re-enrolled, the subject must be re-consented.
3. Age and Reproductive Status

   * Men and women, > or = to 18 years of age
   * Women of childbearing potential (WOCBP) must use method(s) of contraception. WOCBP should therefore use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for Nivolumab to undergo five half lives) after the last dose of investigational drug.
   * Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
   * Women must not be breastfeeding
   * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1 percent per year. Men that are sexually active with WOCBP must follow instructions for birth control when the half life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half lives. The half life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. Given the blinded nature of the study, men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half lives) after the last dose of investigational drug.
   * Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile and azoospermic men do not require contraception.

Exclusion Criteria:

1. Target Disease Exceptions

   * Active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if these have been treated and there is no magnetic resonance imaging (MRI except where contraindicated in which CT scan is acceptable) evidence of progression for at least 8 weeks after treatment is complete and within 28 days prior to first dose of study drug administration. Cases should be discussed with the medical monitor. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
2. Medical History and Concurrent Diseases

   * Prior combination treatment directed against the PD-1/PDL1 (Programmed Death Ligand 1) axis (anti PD 1, anti PD-L1, anti PD L2), and anti CTLA 4 antibody. Prior monotherapy with these agents or other immune-stimulating/regulating agents is permitted.
   * Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
   * Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
   * Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
   * Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
3. Physical and Laboratory Test Findings

   * Any positive test result for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
   * Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
4. Allergies and Adverse Drug Reaction

   * History of allergy to study drug components.
   * History of severe hypersensitivity reaction to any monoclonal antibody.
5. Sex and Reproductive Status

   * WOCBP who are pregnant or breastfeeding
   * Women with a positive pregnancy test at enrolment or prior to administration of study medication.
6. Other Exclusion Criteria

   * Prisoners or subjects who are involuntarily incarcerated
   * Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
To determine the clinical efficacy of the combination treatment of ipilimumab with nivolumab in rare cancers. | at 12 weeks following randomisation then every 6 weeks until disease progression
  Clinical benefit rate for whole population (CR (complete response)+PR (partial response)+SD (stable disease)>3 months)

SECONDARY OUTCOMES:
To identify whether a common predictive biomarker or immune signature can be identified in responding patients that can occur irrespective of tumour type. | Pre-dose samples will be collected during the first two cycles (6 weeks/cycle)
  Pre-dose Blood and Serum samples on Day 1 week 1 and Day 1 week 4 for cycle 1 and Day 1 week 1 for cycle 2 (each cycle is 6 weeks). Optional tumour biopsies will be assessed at Day 1 week 1 and Day 1 week 4 for both cycles 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Study Chair — ONJCRI and Austin Health; Jonathan Cebon, MD, Study Chair — ONJCRI and Austin Health
Locations (5):
- Australia (5):
  - Border Medical Oncology Unit, Albury, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Derived] Klein O, Kee D, Nagrial A, Markman B, Underhill C, Michael M, Jackett L, Lum C, Behren A, Palmer J, Tebbutt NC, Carlino MS, Cebon J. Evaluation of Combination Nivolumab and Ipilimumab Immunotherapy in Patients With Advanced Biliary Tract Cancers: Subgroup Analysis of a Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1405-1409. doi: 10.1001/jamaoncol.2020.2814. PMID 32729929